CLINICAL TRIAL: NCT02348528
Title: A Multi-center, Open-label Extended Access Program of Lenalidomide Plus Low-dose Dexamethasone in Chinese Subjects With Relapsed/Refactory Multiple Myeloma Who Participated in Study CC-5013-MM-021 for at Least One Year.
Brief Title: Open-label Extended Access Program on Lenalidomide Plus Dexamethasone in Chinese Subjects With Relapsed/Refractory Multiple Myeloma Who Participated in CC-5013-MM021 for at Least 1 Year
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-024
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Lenalidomide; Dexamethasone; open-label; CC-5013-MM-021
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and dexamethasone (Experimental): Cycle 1: 25 mg oral lenalidomide once daily on Days 1-21 every 28 Days and 40 mg oral dexamethasone on Days 8, 15, and 22. Cycle 2 and beyond: 25 oral lenalidomide once daily on Days 1-21 every 28 days and 40 mg oral dexamethasone once daily on Days 1, 8, 15, and 22.
  The starting doses of Rd regimen will be the same last doses that the subjects received in Study CC-5013-MM-021, unless event(s) that require dose adjustments (dose modifications, reductions and interruptions) per protocol occurred prior to roll-over.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
CC5013-MM024 is a multicenter, open-label, Extended Access Program (EAP) of lenalidomide plus low dose dexamethasone regimen in Chinese subjects with relapsed or refractory MM who participated in Study CC-5013-MM-021. For subjects who remained progression free under Rd treatment of Study CC-5013-MM-02 1, this LAP offers the option to continue lenalidomide treatment for subjects who have shown therapeutic benefit.

DETAILED DESCRIPTION:
After subjects who are still on treatment have completed at least 1 year of therapy in Study CC-5013-MM-021 (from the start date of lenalidomide treatment), the EAP will allow consented subjects who (1) have remained progression free under Rd treatment in Study CC-SO I3-MM-02 I to roll over to the Treatment Phase of the LAP to continue Rd treatment, and (2) have discontinued Rd therapy and are currently in the Long-Term Follow-up Phase in Study CC-5013-MM-021 to roll over to the Safety Follow-up Phase of the EAP for survival and SPM outcomes. The maximum duration of this LAP program is at least 5 years from the time the last on-study

ELIGIBILITY:
Inclusion Criteria:

Subjects who discontinued treatment but remained for long-term follow-up in the CC-5013-MM-021 study are required to sign an informed consent document (ICD) to roll over to the Safety Follow-up Phase of the Extended Access Program (EAP). These subjects do not require screening for eligibility but must agree to be followed for survival and Second Primary Malignancy (SPM) at a minimum of every 4 months (± 7 days) intervals for at least 5 years from the time the last on-study subject enrolled in Study CC-5013-MM-021.

Subjects who are consented for the Treatment Phase of the EAP must meet the following criteria to continue the same therapy as they received in the Study CC-5013-MM-021:

1. Completed at least 1year of lenalidomide plus low-dose dexamethasone (Rd) treatment and remained progression free under Rd treatment in Study CC-5013-MM-021 at the time of screening visit of this EAP.
2. Able to adhere study visit schedule, compliance with study drug and other protocol requirements in Study CC-5013-MM-024.
3. Consented to the EAP protocol.
4. Must agree to comply with all Pregnancy Prevention requirements.
5. Females of childbearing potential (FCBP)1:

   * Must agree to use, and be able to comply with, at least 2 forms of reliable contraception simultaneously or to practice complete abstinence from heterosexual intercourse without interruption, from transferring/rolling over from the CC-5013-MM-021 study, at the screening visit for eligibility, throughout study drug therapy (including dose interruptions) and for 28 days after the end of study drug therapy, even if she has amenorrhea. This applies even if the subject practices complete and continued abstinence confirmed on a monthly basis.
   * Must agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 IU/mL (i.e., negative pregnancy test) at screening for eligibility and then every 28 days while on study. For any FCBP, pregnancy testing must continue at the same frequency as during the MM-021 study. If regular or no menstrual cycles, she must agree to ongoing pregnancy testing during the course of the study (every 28 days), during dose interruptions, at study discontinuation and 28 days following study drug discontinuation. If menstrual cycles are irregular, pregnancy testing must occur every 14 days while on study, at study discontinuation and at 14 and 28 days following study drug discontinuation. This requirement also applies to females of childbearing potential who practice complete and continued sexual abstinence.
   * Must agree not to breastfeed during study drug therapy and for at least 28 days following study drug discontinuation.
6. Male subjects:

   * Must agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and at least 28 days following study drug discontinuation.
   * Must agree to not donate semen or sperm during study drug therapy and for at least 28 days following study drug discontinuation.

Subjects who have a positive finding of pregnancy testing at screening will not be eligible for the Treatment Phase of the EAP but will be consented for the Safety Follow-up Phase in the EAP.

Exclusion Criteria:

* Subjects will not continue treatment at the discretion of the physician if any of the following criteria occurred during treatment in the CC-5013-MM-021 study or during the Screening Phase.

All subjects that are not eligible to continue treatment will enter the Safety Follow-up Phase:

1. Serious hypersensitivity or anaphylaxis to lenalidomide or dexamethasone.
2. Serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document.
3. Any other condition, including the presence of serious laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Previously discontinued lenalidomide treatment due to toxicity.
5. Newly diagnosed malignancy other than Multiple Myeloma (MM), except the following:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system) or prostate cancer that is curative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | approximately 4 years
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. A diagnosis or syndrome should be recorded on the AE page of the electronic case report form (eCRF) rather than the individual signs or symptoms of the diagnosis or syndrome. An overdose, accidental or intentional, whether or not it is associated with an AE, or abuse, withdrawal, sensitivity or toxicity to an investigational product should be reported as an AE. If an overdose is associated with an AE, the overdose and adverse event should be reported as separate terms.

SECONDARY OUTCOMES:
Progression Free Survival (PFS | approximately 4 years
  Progression Free Survival is defined as the time between randomization and the first documented progressive disease or death, whichever occurred first
Time to Progression (TTP) | approximately 4 years
  Time to progression is defined as the time between randomization and disease progression as determined by the investigator
Overall Survival (OS) | approximately 4 years
  Overall Survival is defined as the time between randomization and death Safety Issue: No
  Click here to enter additional Secondary Outcome Measures following the format above.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jacques, MD, Study Director — Celgene Corporation
Locations (10):
- China (10):
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The 301 Hospital-Chinese PLA General Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Guangdong General Hospital, Guangzhou
  - Nanfang Hospital of Southern medicine university in Guangzhou, Guangzhou
  - 1st Hospital Zhejiang University (The First Affiliated Hospital of Zhejiang University ), Hangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai 6th Hospital, Shanghai
  - The 1st Hospital of Soochow University, Suzhou

REFERENCES:
- [Background] Du X, Jin J, Cai Z, Chen F, Zhou DB, Yu L, Ke X, Li X, Wu D, Meng F, DeMarco D, Zhang J, Mei J, Hou J. Long-term use of lenalidomide and low-dose dexamethasone in Chinese patients with relapsed/refractory multiple myeloma: MM-024 Extended Access Program. BMC Cancer. 2016 Jan 28;16:46. doi: 10.1186/s12885-016-2069-8. PMID 26821931
- [Background] Soyer N, Patir P, Uysal A, Duran M, Unal HD, Durusoy R, Tombuloglu M, Sahin F, Tobu M, Vural F, Saydam G. Efficacy and safety of lenalidomide and dexamethasone in patients with relapsed/ refractory multiple myeloma: a real-life experience. Turk J Med Sci. 2018 Aug 16;48(4):777-785. doi: 10.3906/sag-1712-160. PMID 30119153
- [Background] Dinner S, Dunn TJ, Price E, Coutre SE, Gotlib J, Berube C, Kaufman GP, Medeiros BC, Liedtke M. A phase I, open-label, dose-escalation study of amrubicin in combination with lenalidomide and weekly dexamethasone in previously treated adults with relapsed or refractory multiple myeloma. Int J Hematol. 2018 Sep;108(3):267-273. doi: 10.1007/s12185-018-2468-5. Epub 2018 May 25. PMID 29802551
- [Background] Lund J, Gruber A, Lauri B, Duru AD, Blimark C, Swedin A, Hansson M, Forsberg K, Ahlberg L, Carlsson C, Waage A, Gimsing P, Vangsted AJ, Frolund U, Holmberg E, Gahrton G, Alici E, Hardling M, Mellqvist UH, Nahi H. Lenalidomide versus lenalidomide + dexamethasone prolonged treatment after second-line lenalidomide + dexamethasone induction in multiple myeloma. Cancer Med. 2018 Jun;7(6):2256-2268. doi: 10.1002/cam4.1422. Epub 2018 Apr 19. PMID 29673108
- [Background] Dimopoulos MA, Lonial S, Betts KA, Chen C, Zichlin ML, Brun A, Signorovitch JE, Makenbaeva D, Mekan S, Sy O, Weisel K, Richardson PG. Elotuzumab plus lenalidomide and dexamethasone in relapsed/refractory multiple myeloma: Extended 4-year follow-up and analysis of relative progression-free survival from the randomized ELOQUENT-2 trial. Cancer. 2018 Oct 15;124(20):4032-4043. doi: 10.1002/cncr.31680. Epub 2018 Sep 11. PMID 30204239
- [Background] Cella D, McKendrick J, Kudlac A, Palumbo A, Oukessou A, Vij R, Zyczynski T, Davis C. Impact of elotuzumab treatment on pain and health-related quality of life in patients with relapsed or refractory multiple myeloma: results from the ELOQUENT-2 study. Ann Hematol. 2018 Dec;97(12):2455-2463. doi: 10.1007/s00277-018-3469-4. Epub 2018 Sep 4. PMID 30178193
- [Background] Wilke T, Mueller S, Bauer S, Pitura S, Probst L, Ratsch BA, Salwender H. Treatment of relapsed refractory multiple myeloma: which new PI-based combination treatments do patients prefer? Patient Prefer Adherence. 2018 Nov 9;12:2387-2396. doi: 10.2147/PPA.S183187. eCollection 2018. PMID 30519004
- [Background] Alahmadi M, Masih-Khan E, Atenafu EG, Chen C, Kukreti V, Tiedemann R, Trudel S, Reece DE. Addition of Cyclophosphamide "On Demand" to Lenalidomide and Corticosteroids in Patients With Relapsed/Refractory Multiple Myeloma-A Retrospective Review of a Single-center Experience. Clin Lymphoma Myeloma Leuk. 2019 Apr;19(4):e195-e203. doi: 10.1016/j.clml.2018.12.007. Epub 2018 Dec 20. PMID 30723035
- [Background] Mark TM, Forsberg PA, Rossi AC, Pearse RN, Pekle KA, Perry A, Boyer A, Tegnestam L, Jayabalan D, Coleman M, Niesvizky R. Phase 2 study of clarithromycin, pomalidomide, and dexamethasone in relapsed or refractory multiple myeloma. Blood Adv. 2019 Feb 26;3(4):603-611. doi: 10.1182/bloodadvances.2018028027. PMID 30792190
- [Background] Ailawadhi S, DerSarkissian M, Duh MS, Lafeuille MH, Posner G, Ralston S, Zagadailov E, Ba-Mancini A, Rifkin R. Cost Offsets in the Treatment Journeys of Patients With Relapsed/Refractory Multiple Myeloma. Clin Ther. 2019 Mar;41(3):477-493.e7. doi: 10.1016/j.clinthera.2019.01.009. Epub 2019 Feb 14. PMID 30773308